CLINICAL TRIAL: NCT03872999
Title: Developing a Multi-scale Account of Attentional Control as the Constraining Interface Between Vision and Action (MAC-Brain).
Brief Title: Attentional Control
Acronym: MACBRAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL19_0127; 2019-A00713-54 (Other: ID-RCB)
Record Dates: First submitted 2019-03-08; First posted 2019-03-13 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Attention Control; Healthy Volunteers
Keywords: Attention; Control; Functional Magnetic Resonance Imaging (fMRI); Parietal; Space
MeSH Terms: interventions — Functional Neuroimaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Attentional Control (Experimental): Visuo-spatial attentional tasks with simple stimuli during functional magnetic resonance imaging (fMRI) scanning.
  Interventions: Other: Functional brain imaging without any contrast agent

INTERVENTIONS:
Other: Functional brain imaging without any contrast agent — During the functional magnetic resonance imaging (fMRI) protocol, the subject will perform the attentional task while whole-brain activity will be recorded using Echo Planar Imaging (EPI) that measures the Blood Oxygen Level Dependent (BOLD) signal (2x2x2 isotropic voxels, Echo Time (ET) = 30 ms, Repetition Time (RT) = 2.5 sec). The functional session will be subdivided into several parts ("Runs", duration: 10-15 min). Together with the functional data, the protocol will include a structural scan (T1 weighted, 1x1x1 mm voxels; duration 5-7 min) and a field mapping sequence (duration: 1 min).

SUMMARY:
The project is dedicated to understanding the integration within the brain of signals of different natures that contribute to attentional control. The investigator will make use of standardized experimental displays involving the discrimination of a target (tilted-bar) presented together with 3 distractor items, with one stimulus in each visual quadrant. Across three fMRI experiments in healthy participants, the investigator will manipulate different types of signals that will guide the subject's attention towards one of the four quadrants: Exp 1 - task instruction & item salience; Exp 2 - probabilistic target location; Exp 3 - probabilistic reward. The investigator expects that irrespective of the nature of the control signal, activity in dorsal parietal cortex will index the currently relevant/attended location. Moreover, The investigator expects that upon changes of the most relevant location, one will observe activation of the ventral parietal cortex, plus increased inter-regional connectivity between ventral and dorsal parietal regions - again irrespective of the nature of the attention guiding signals.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 to 40 years old

Exclusion Criteria:

* Previous neurologic or psychiatric disease.
* Cognitive deficits restricting understanding of the tasks.
* Pregnant or breath-feeding women.
* Persons under guardianship, curator or any other administrative or judicial measure of deprivation of rights or liberty.
* Subjects currently participating in other study.

Additional exclusion criteria for a functional magnetic resonance imaging (fMRI) recording:

* Neurologic, cardiac electrostimulation or defibrillator.
* Cardiac prostheses
* Intracranial clips or clamps
* Cerebrospinal fluid disorders
* Metal particles in the eyes
* Metal dental or articular prostheses
* Diffusion pomp or other infusion system
* Claustrophobia
* Head tattoo, make-up, hair gel
* Have any copper intrauterine device

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2019-07-05 (Actual); Primary Completion 2019-07-05 (Actual); Study Completion 2021-06-21 (Actual)

PRIMARY OUTCOMES:
Changes of hemodynamic response in dorsal parietal regions representing specific spatial locations (visual quadrants) | Day 0
  After spatial pre-processing of individual series of functional magnetic resonance imaging (fMRI) scans, normalization and smoothing as suggested for Statistical Parametric Mapping (SPM) analysis, the different attentional conditions will be modeled and convolved with canonical Hemodynamic Response Function (HRF). The model will be estimated according to the algorithm of SPM. Using a Region of Interest (ROI) approach, the investigator will extract the signal in dorsal parietal regions representing the four visual quadrants, and will compare activity as a function of the attended / most relevant location. The main hypothesis will be confirmed by activation of the ROI corresponding to the currently attended location, irrespective of the nature of the signal guiding attention (i.e. common effects in Exp 1-3).

SECONDARY OUTCOMES:
Evaluation of the brain hemodynamic response | Day 0
  The investigator will search for relations between changes over time of the most relevant location (trial history) and the re-organization of attentional representations by investigating the activity and connectivity of the ventral parietal cortex. For this, the investigator will model events corresponding to changes in attention location and test for local activation of the ventral parietal cortex, as well as changes in connectivity (correlation) between ventral and dorsal parietal regions. The secondary hypothesis will be confirmed by increased activation in ventral parietal cortex, plus increased connectivity between ventral and dorsal parietal regions, at the time of a change of the most relevant location, irrespective of the nature of the signal guiding attention (i.e. common effects in Exp 1-3).
Evaluation of the connectivity of the ventral parietal cortex at the time when there is a change of the most relevant spatial location/visual quadrant. x² | Day 0
  The investigator will search for relations between changes over time of the most relevant location (trial history) and the re-organization of attentional representations by investigating the activity and connectivity of the ventral parietal cortex. For this, the investigator will model events corresponding to changes in attention location, and test for local activation of the ventral parietal cortex, as well as changes of connectivity (correlation) between ventral and dorsal parietal regions. The secondary hypothesis will be confirmed by increased activation in ventral parietal cortex, plus increased connectivity between ventral and dorsal parietal regions, at the time of a change of the most relevant location, irrespective of the nature of the signal guiding attention (i.e. common effects in Exp 1-3).

CONTACTS AND LOCATIONS:
Overall Officials: Emiliano Macaluso, Prof., Principal Investigator — INSERM U1028 - Equipe ImpAct CRNL
Locations (1):
- Inserm U1028 Equipe Impact, Bron, France